CLINICAL TRIAL: NCT05315297
Title: Pulsed Electromagnetic Field (PEMF) Therapy in Thumb CMC Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Raymond Chou, Clinical Assistant Professor of Orthopaedic Surgery, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 64143
Record Dates: First submitted 2022-03-15; First posted 2022-04-07 (Actual); Results first posted 2025-07-24 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Thumb Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- PEMF device (Experimental)
  Interventions: Device: PEMF device
- Sham PEMF device (Sham Comparator)
  Interventions: Device: Sham PEMF device

INTERVENTIONS:
Device: PEMF device — PEMF device wear overnight daily for four weeks
  Other Names: ActiPatch
  Arms: PEMF device
Device: Sham PEMF device — Sham PEMF device wear overnight daily for four weeks. Sham PEMF devices do not emit a radiofrequency electromagnetic field but are otherwise identical in appearance to the PEMF device
  Arms: Sham PEMF device

SUMMARY:
Long-Term Objective: Determine if high-frequency PEMF therapy reduces pain in patients with thumb carpometacarpal (CMC) joint osteoarthritis (OA).

Study Design and Methods: This will be a randomized controlled pilot study with 60 subjects with CMC OA randomly divided in two groups. Thirty subjects will receive high-frequency PEMF therapy overlying the CMC joint overnight daily for four weeks. The other 30 subjects will receive a sham PEMF therapy device applied to the same joint overnight daily for four weeks. Pain and function questionnaires will be obtained for all patients at enrollment, four weeks, and six weeks.

ELIGIBILITY:
Inclusion Criteria:

* an existing diagnosis of CMC OA by a hand specialist based on clinically (tenderness to palpation at the CMC joint and/or positive CMC grind test) and/or radiographically identified CMC OA
* reported pain intensity during activities of daily living less than 7 on the Numeric Pain Rating Scale (NPRS)

Exclusion Criteria:

* pregnant
* unable to consent
* with current infection in hand or upper extremity
* have had prior fracture, significant hand injury, tenosynovitis, complex regional pain syndrome, and/or Dupuytren's disease affecting the thumb
* history of surgical or procedural intervention for CMC OA in the hand of study interest
* do not speak English
* have hand or wrist implants
* have heart or brain implants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2023-06-20 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Chou, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Medicine Outpatient Center, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PEMF Device | Sham PEMF Device
Started | 31 | 30
Completed 4 Weeks | 26 | 28
Completed | 25 | 25
Not Completed | 6 | 5
Not completed — Lost to Follow-up | 6 | 4
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PEMF Device | Sham PEMF Device | Total
Number analyzed (Participants) | 31 | 30 | 61
Age, Continuous [Median (Full Range); unit: years] | 67 [40 to 82] | 65 [40 to 78] | 66 [40 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 25 | 46
  Male | 10 | 5 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 31 | 30 | 61
Numeric Pain Rating Scale (NPRS) [Median (Full Range); unit: units on a scale] — NPRS is a unidimensional measure of pain intensity in adults. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
  units on a scale | 5 [4 to 7] | 5 [2 to 7] | 5 [2 to 7]
Patient Rated Wrist/Hand Evaluation (PRWHE) [Median (Full Range); unit: score on a scale] — PRWHE consists of 15 questions on symptoms with daily activities scored on a 11-point numeric scale, in which '0' represents no difficulty or pain. The total score is then scaled from '0' representing no disability to '100' representing most severe disability.
  score on a scale | 47 [30 to 85] | 48 [25 to 91] | 48 [25 to 91]
Single Assessment Numeric Evaluation (SANE) [Median (Full Range); unit: units on a scale] — SANE is a single-question outcome measure that asks patient to rate their function of the treated area on a scale from '0' to '100' ("For the problem that you are seeking treatment for today, out of 100% (100% being normal), how would you rate the function of your RIGHT/LEFT thumb today?").
  units on a scale | 70 [40 to 90] | 65 [10 to 90] | 65 [10 to 90]

OUTCOME MEASURES:

1. Primary Outcome: Numeric Pain Rating Scale (NPRS)
Description: NPRS is a unidimensional measure of pain intensity in adults. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
Time Frame: 4 weeks
Population: Excludes participants with missing data
Measure: Median (Full Range); unit: units on a scale
Arm/Group | PEMF Device | Sham PEMF Device
Number analyzed (Participants) | 25 | 26
units on a scale | 3 [0 to 7] | 3 [1 to 9]
Statistical Analysis 1: Comparison: PEMF Device vs Sham PEMF Device; Test type: Superiority; p = 0.87, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Numeric Pain Rating Scale (NPRS)
Description: as for outcome 1
Time Frame: 6 weeks
Population: Excludes participants with missing data
Measure: Median (Full Range); unit: units on a scale
Arm/Group | PEMF Device | Sham PEMF Device
Number analyzed (Participants) | 25 | 25
units on a scale | 3 [1 to 6] | 4 [1 to 7]
Statistical Analysis 1: Comparison: PEMF Device vs Sham PEMF Device; Test type: Superiority; p = 0.13, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Patient-Rated Wrist/Hand Evaluation (PRWHE)
Description: PRWHE consists of 15 questions on symptoms with daily activities scored on a 11-point numeric scale, in which '0' represents no difficulty or pain. The total score is then scaled from '0' representing no disability to '100' representing most severe disability.
Time Frame: 4 weeks
Population: Excludes participants with missing data
Measure: Median (Full Range); unit: score on a scale
Arm/Group | PEMF Device | Sham PEMF Device
Number analyzed (Participants) | 25 | 26
score on a scale | 39 [5 to 70] | 39 [5 to 83]
Statistical Analysis 1: Comparison: PEMF Device vs Sham PEMF Device; Test type: Superiority; p = 0.78, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Single Assessment Numeric Evaluation (SANE)
Description: SANE is a single-question outcome measure that asks patient to rate their function of the treated area on a scale from '0' to '100' ("For the problem that you are seeking treatment for today, out of 100% (100% being normal), how would you rate the function of your RIGHT/LEFT thumb today?").
Time Frame: 4 weeks
Population: Excludes participants with missing data
Measure: Median (Full Range); unit: units on a scale
Arm/Group | PEMF Device | Sham PEMF Device
Number analyzed (Participants) | 22 | 22
units on a scale | 75 [40 to 100] | 75 [20 to 98]
Statistical Analysis 1: Comparison: PEMF Device vs Sham PEMF Device; Test type: Superiority; p = 0.59, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Patient-Rated Wrist/Hand Evaluation (PRWHE)
Description: as for outcome 3
Time Frame: 6 weeks
Population: Excludes participants with missing data
Measure: Median (Full Range); unit: score on a scale
Arm/Group | PEMF Device | Sham PEMF Device
Number analyzed (Participants) | 25 | 25
score on a scale | 35 [12 to 66] | 43 [9 to 88]
Statistical Analysis 1: Comparison: PEMF Device vs Sham PEMF Device; Test type: Superiority; p = 0.37, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Single Assessment Numeric Evaluation (SANE)
Description: as for outcome 4
Time Frame: 6 weeks
Population: Excludes participants with missing data
Measure: Median (Full Range); unit: units on a scale
Arm/Group | PEMF Device | Sham PEMF Device
Number analyzed (Participants) | 22 | 23
units on a scale | 73 [30 to 100] | 65 [20 to 99]
Statistical Analysis 1: Comparison: PEMF Device vs Sham PEMF Device; Test type: Superiority; p = 0.19, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Data collected weekly for 6 weeks
Arm/Group | PEMF Device | Sham PEMF Device
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/30
Other Adverse Events (participants affected / at risk) | 5/31 | 4/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PEMF Device (N=31) | Sham PEMF Device (N=30)
Skin allergy/blistering (Skin and subcutaneous tissue disorders) | 3 | 2 — Attributed to the adhesive tape used to secure the device
Increased thumb pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Increased Dupuytren's contracture (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-06): https://cdn.clinicaltrials.gov/large-docs/97/NCT05315297/Prot_SAP_000.pdf